CLINICAL TRIAL: NCT04202354
Title: A Phase 1/2a Single and Multiple Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of ARO-HSD in Normal Healthy Volunteers as Well as in Patients With NASH or Suspected NASH
Brief Title: Study of ARO-HSD in Healthy Volunteers and Patients With Non-Alcoholic Steatohepatitis (NASH) or Suspected NASH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROHSD1001
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Cohort 1: ARO-HSD 25 mg (Experimental): Normal healthy volunteers randomized to double blind ARO-HSD 25 mg on Day 1 only.
  Interventions: Drug: ARO-HSD Injection
- Cohort 1: Placebo (Placebo Comparator): Normal healthy volunteers randomized to double blind placebo on Day 1 only.
  Interventions: Drug: sterile normal saline (0.9% NaCl)
- Cohort 2: ARO-HSD 50 mg (Experimental): Normal healthy volunteers randomized to double blind ARO-HSD 50 mg on Day 1 only.
  Interventions: Drug: ARO-HSD Injection
- Cohort 2: Placebo (Placebo Comparator): Normal healthy volunteers randomized to double blind placebo on Day 1 only.
  Interventions: Drug: sterile normal saline (0.9% NaCl)
- Cohort 3: ARO-HSD 100 mg (Experimental): Normal healthy volunteers randomized to double blind ARO-HSD 100 mg on Day 1 only.
  Interventions: Drug: ARO-HSD Injection
- Cohort 3: Placebo (Placebo Comparator): Normal healthy volunteers randomized to double blind placebo on Day 1 only.
  Interventions: Drug: sterile normal saline (0.9% NaCl)
- Cohort 4: ARO-HSD 200 mg (Experimental): Normal healthy volunteers randomized to double blind ARO-HSD 200 mg on Day 1 only.
  Interventions: Drug: ARO-HSD Injection
- Cohort 4: Placebo (Placebo Comparator): Normal healthy volunteers randomized to double blind placebo on Day 1 only.
  Interventions: Drug: sterile normal saline (0.9% NaCl)
- Cohort 1b: ARO-HSD 25 mg (Experimental): Participants with suspected non-alcoholic steatohepatitis (NASH) receive open-label ARO-HSD 25 mg on Days 1 and 29.
  Interventions: Drug: ARO-HSD Injection
- Cohort 3b: ARO-HSD 100 mg (Experimental): Participants with suspected NASH receive open-label ARO-HSD 100 mg on Days 1 and 29.
  Interventions: Drug: ARO-HSD Injection
- Cohort 4b: ARO-HSD 200 mg (Experimental): Participants with suspected NASH receive open-label ARO-HSD 200 mg on Days 1 and 29.
  Interventions: Drug: ARO-HSD Injection

INTERVENTIONS:
Drug: ARO-HSD Injection — single or multiple doses of ARO-HSD by subcutaneous (sc) injections
  Arms: Cohort 1: ARO-HSD 25 mg; Cohort 1b: ARO-HSD 25 mg; Cohort 2: ARO-HSD 50 mg; Cohort 3: ARO-HSD 100 mg; Cohort 3b: ARO-HSD 100 mg; Cohort 4: ARO-HSD 200 mg; Cohort 4b: ARO-HSD 200 mg
Drug: sterile normal saline (0.9% NaCl) — calculated volume to match active treatment, by sc injection
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics of single and multiple doses of ARO-HSD in healthy adult volunteers and in patients with NASH or suspected NASH.

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* On a stable diet for at least 4 weeks with no plans to significantly alter diet or weight over course of study
* Normal electrocardiogram (ECG) at Screening
* No abnormal finding of clinical relevance (other than NASH, suspected NASH in patients) at Screening that could adversely impact subject safety during the study or adversely impact study results.

Exclusion Criteria:

* Clinically significant health concerns (other than NASH, suspected NASH in patients)
* Human immunodeficiency virus (HIV) infection, seropositive for Hepatitis B Virus (HBV), seropositive for Hepatitis C Virus (HCV)
* Uncontrolled hypertension
* Excessive use of alcohol within three months prior to Screening
* Use of illicit drugs within 1 year prior to Screening, or positive urine drug screen at Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study

NOTE: additional inclusion/exclusion criteria may apply, per protocol

-

-

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland Clinical Studies, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mak LY, Gane E, Schwabe C, Yoon KT, Heo J, Scott R, Lee JH, Lee JI, Kweon YO, Weltman M, Harrison SA, Neuschwander-Tetri BA, Cusi K, Loomba R, Given BD, Christianson DR, Garcia-Medel E, Yi M, Hamilton J, Yuen MF. A phase I/II study of ARO-HSD, an RNA interference therapeutic, for the treatment of non-alcoholic steatohepatitis. J Hepatol. 2023 Apr;78(4):684-692. doi: 10.1016/j.jhep.2022.11.025. Epub 2022 Dec 10. PMID 36513186

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following Screening, Cohorts 1 through 4 (normal healthy volunteers) enrolled eligible participants, randomly assigned 1:1 to receive a single subcutaneous (SC) dose of ARO-HSD or placebo on Day 1. Per protocol, the placebo cohorts were pooled for data analysis.
Groups:
- Cohorts 1-4: Pooled Placebo: Normal healthy volunteers randomized to double blind placebo on Day 1 only.
- Cohort 4b: ARO-HSD 200 mg: Participants with suspected NASH received open-label ARO-HSD 200 mg on Days 1 and 29.
Period: Overall Study
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg | Cohorts 1-4: Pooled Placebo | Cohort 1b: ARO-HSD 25 mg | Cohort 3b: ARO-HSD 100 mg | Cohort 4b: ARO-HSD 200 mg
Started | 4 | 4 | 4 | 4 | 16 | 6 | 6 | 6
Completed | 4 | 4 | 4 | 4 | 16 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1b: ARO-HSD 25 mg: Participants with suspected NASH receive open-label ARO-HSD 25 mg on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg | Cohorts 1-4: Pooled Placebo | Cohort 1b: ARO-HSD 25 mg | Cohort 3b: ARO-HSD 100 mg | Cohort 4b: ARO-HSD 200 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16 | 6 | 6 | 6 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 16 | 6 | 6 | 6 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 10 | 1 | 1 | 2 | 21
  Male | 3 | 2 | 3 | 1 | 6 | 5 | 5 | 4 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 1 | 1 | 4 | 5 | 4 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 2 | 2 | 11 | 2 | 0 | 1 | 23
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 3 | 2 | 4 | 16 | 6 | 6 | 6 | 47
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Possibly or Probably Related to Treatment
Description: Adverse event (AE)=any untoward medical occurrence that does not necessarily have to have a causal relationship with this treatment. TEAEs=AEs with onset after administration of the study drug, or when a pre-existing medical condition increases in severity or frequency after study drug administration. Serious adverse event (SAE)= an AE that results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event or reaction.
Time Frame: From first dose of study drug through Day 113 (±5 days)
Population: Safety Population: all enrolled participants who received at least one dose of active drug or placebo.
Measure: Number; unit: participants
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg | Cohorts 1-4: Pooled Placebo | Cohort 1b: ARO-HSD 25 mg | Cohort 3b: ARO-HSD 100 mg | Cohort 4b: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16 | 6 | 6 | 6
participants | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 2

2. Secondary Outcome: Pharmacokinetics (PK) of ARO-HSD: Plasma Concentrations
Time Frame: Normal Healthy Volunteers: Day 1: 2 hours pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 8, 12, 18, 24; Day 2: 48 hours post-dose, Days 8, 15, 29. NASH Participants: Day 1: 2 hours pre-dose, 30 minutes, 1, 2, 24, hours post-dose, Days 8, 15, 29
Population: PK Analysis Set: all participants who received at least one dose of active study treatment and had sufficient plasma concentration data to characterize PK profile. Participants with sufficient data at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg | Cohort 1b: ARO-HSD 25 mg | Cohort 3b: ARO-HSD 100 mg | Cohort 4b: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 6 | 6
ng/mL
  2 hours pre-dose | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000)
  15 minutes post-dose: number analyzed (Participants) | 4 | 3 | 4 | 4 | 0 | 0 | 0
  15 minutes post-dose | 56.7555 (13.2117) | 60.7480 (52.6374) | 101.4768 (66.7517) | 275.6855 (261.1693) |  |  |
  30 minutes post-dose: number analyzed (Participants) | 4 | 4 | 4 | 4 | 6 | 5 | 6
  30 minutes post-dose | 67.6780 (13.9394) | 116.6108 (70.4360) | 160.9810 (72.2119) | 445.7370 (316.1025) | 22.13370 (8.3169) | 123.2292 (11.5639) | 174.1368 (127.8926)
  1 hour post-dose | 66.6098 (14.6623) | 134.8668 (66.4452) | 211.1088 (78.3225) | 531.6415 (213.0969) | 29.3950 (8.2373) | 158.0703 (36.7514) | 251.3230 (133.5201)
  2 hours post-dose: number analyzed (Participants) | 4 | 4 | 4 | 3 | 6 | 6 | 6
  2 hours post-dose | 53.5845 (9.4115) | 137.1443 (53.1775) | 219.4920 (108.8893) | 510.3820 (146.3129) | 26.4290 (7.2923) | 166.2240 (45.4507) | 286.9603 (103.4747)
  4 hours post-dose: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 0 | 0
  4 hours post-dose | 60.8553 (4.2935) | 157.5515 (64.5494) | 253.6468 (91.5590) | 542.9808 (80.1204) |  |  |
  8 hours post-dose: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 0 | 0
  8 hours post-dose | 53.9558 (12.2129) | 136.8678 (49.6823) | 255.7058 (27.2111) | 534.2020 (56.0211) |  |  |
  12 hours post-dose: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 0 | 0
  12 hours post-dose | 33.7875 (6.5592) | 80.2873 (26.8625) | 180.7433 (54.0979) | 363.3568 (35.9755) |  |  |
  18 hours post-dose: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 0 | 0
  18 hours post-dose | 12.5088 (5.5194) | 17.7438 (12.6477) | 75.3893 (32.1815) | 176.4455 (41.8914) |  |  |
  24 hours post-dose | 2.0123 (1.7888) | 2.9088 (2.3774) | 20.6793 (12.8362) | 65.4435 (28.6583) | 6.7428 (4.3051) | 25.5277 (9.0820) | 84.2982 (28.8905)
  48 hours post-dose: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 0 | 0
  48 hours post-dose | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 1.8418 (1.2854) |  |  |
  Day 8: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 5 | 4
  Day 8 | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) |  | 0.0000 (0.0000) | 0.0000 (0.0000)
  Day 15: number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 6 | 6
  Day 15 | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000)
  Day 29: number analyzed (Participants) | 0 | 4 | 4 | 3 | 6 | 6 | 6
  Day 29 |  | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000)

3. Secondary Outcome: PK of ARO-HSD in Normal Healthy Volunteers: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: PK Analysis Set: all participants who received at least one dose of active study treatment and had sufficient plasma concentration data to characterize PK profile. Normal healthy volunteer cohorts only.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
ng/mL | 74.0 (11.5) | 184 (52.2) | 294 (60.3) | 644 (183)

4. Secondary Outcome: PK of ARO-HSD in Normal Healthy Volunteers: Time to Reach Cmax (Tmax)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hours | 2.5 [0.5 to 8.0] | 3.0 [0.5 to 8.0] | 8.0 [4.0 to 8.0] | 3.0 [0.5 to 8.0]

5. Secondary Outcome: PK of ARO-HSD in Normal Healthy Volunteers: Terminal Elimination Half-Life (t1/2)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hours | 3.3 (0.90) | 2.5 (0.6) | 3.7 (0.9) | 4.5 (0.7)

6. Secondary Outcome: PK of ARO-HSD in Normal Healthy Volunteers: Area Under the Concentration-Time Curve From Dosing (Time 0) to the Time of the Last Measured Concentration (AUClast)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
h*ng/mL | 788 (43.5) | 1830 (346) | 3670 (549) | 8450 (479)

7. Secondary Outcome: PK of ARO-HSD in Normal Healthy Volunteers: Area Under the Curve From Time 0 to Infinity (AUCinf)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
h*ng/mL | 806 (38.4) | 1840 (343) | 3790 (587) | 8500 (506)

8. Secondary Outcome: Secondary: PK of ARO-HSD in Normal Healthy Volunteers: Oral Clearance (CL/F)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
L/hour | 31.1 (1.48) | 27.9 (4.96) | 26.8 (3.65) | 23.6 (1.43)

9. Secondary Outcome: PK of ARO-HSD in Normal Healthy Volunteers: Apparent Volume of Distribution During the Terminal-Phase (Vz/F)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24, 48 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
L | 148 (38.7) | 99.9 (29.3) | 141 (37.6) | 153 (27.7)

10. Secondary Outcome: Urine PK of ARO-HSD in Normal Healthy Volunteers: Amount of Unchanged Drug Recovered in Urine Over 0-24 Hours Postdose (Ae0-24h)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
mg | 1.56 (0.12) | 3.64 (0.75) | 6.67 (3.21) | 45.8 (9.66)

11. Secondary Outcome: Urine PK of ARO-HSD in Normal Healthy Volunteers: Percentage of the Administrated Drug Recovered in Urine Over 0-24 Hours (Fe0-24h)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of study drug
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
percentage of study drug | 6.23 (0.47) | 7.29 (1.50) | 6.67 (3.21) | 22.9 (4.83)

12. Secondary Outcome: Urine PK of ARO-HSD in Normal Healthy Volunteers: Renal Clearance (CLr)
Time Frame: Day 1: Predose, 15 minutes, 30 minutes, 1, 2, 4, 8 12, 18, 24 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
L/hour | 1.97 (0.14) | 1.99 (0.17) | 1.82 (0.88) | 5.75 (1.43)

ADVERSE EVENTS:
Time Frame: Screening through Day 113 (±5 days)
Groups:
- Cohort 3: ARO-HSD 100 mg: Normal healthy volunteers randomized to double blind ARO-HSD 200 mg on Day 1 only.
- Cohort 4: ARO-HSD 200 mg: Normal healthy volunteers randomized to double blind ARO-HSD ≤ 200 mg on Day 1 only
Arm/Group | Cohort 1: ARO-HSD 25 mg | Cohort 2: ARO-HSD 50 mg | Cohort 3: ARO-HSD 100 mg | Cohort 4: ARO-HSD 200 mg | Cohorts 1-4: Pooled Placebo | Cohort 1b: ARO-HSD 25 mg | Cohort 3b: ARO-HSD 100 mg | Cohort 4b: ARO-HSD 200 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/16 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/16 | 0/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 4/4 | 1/4 | 4/4 | 3/4 | 10/16 | 3/6 | 2/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ARO-HSD 25 mg (N=4) | Cohort 2: ARO-HSD 50 mg (N=4) | Cohort 3: ARO-HSD 100 mg (N=4) | Cohort 4: ARO-HSD 200 mg (N=4) | Cohorts 1-4: Pooled Placebo (N=16) | Cohort 1b: ARO-HSD 25 mg (N=6) | Cohort 3b: ARO-HSD 100 mg (N=6) | Cohort 4b: ARO-HSD 200 mg (N=6)
Soft tissue injury (Injury, poisoning and procedural complications) | NA | NA | NA | NA | NA | NA | NA | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ARO-HSD 25 mg (N=4) | Cohort 2: ARO-HSD 50 mg (N=4) | Cohort 3: ARO-HSD 100 mg (N=4) | Cohort 4: ARO-HSD 200 mg (N=4) | Cohorts 1-4: Pooled Placebo (N=16) | Cohort 1b: ARO-HSD 25 mg (N=6) | Cohort 3b: ARO-HSD 100 mg (N=6) | Cohort 4b: ARO-HSD 200 mg (N=6)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Morning sickness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04202354/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04202354/SAP_001.pdf